CLINICAL TRIAL: NCT05810740
Title: A Randomized, Single-center, Open-label, Single Dose, Two-period, Crossover Pivotal Bioequivalence Study Comparing Binimetinib 3 x 15 mg and 45 mg Tablets in Healthy Participants
Brief Title: Bioequivalence Binimetinib 3 x 15 mg and 45 mg Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: W00074CI103_1PF74
Record Dates: First submitted 2022-07-22; First posted 2023-04-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Melanoma; BRAF V600 Mutation; Unresectable Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binimetinib 15 mg then Binimetinib 45 mg (Experimental): Participants first received a single dose of 3 tablets of Binimetinib 15 mg orally in fasted conditions in the morning on day 1 of a 5-day period. After a washout period of 7 days, they then received a single dose of 1 tablet of Binimetinib 45 mg orally in fasted conditions in the morning for five days on day 1 of a second 5-day period.
  Interventions: Drug: Binimetinib 15 MG; Drug: Binimetinib 45 MG
- Binimetinib 45 mg then Binimetinib 15 mg (Experimental): Participants first received a single dose of 1 tablet of Binimetinib 45 mg orally in fasted conditions in the morning on day 1 of a 5-day period. After a washout period of 7 days, they then received a single dose of 3 tablets of Binimetinib 15 mg orally in fasted conditions in the morning for five days on day 1 of a second 5-day period.
  Interventions: Drug: Binimetinib 15 MG; Drug: Binimetinib 45 MG

INTERVENTIONS:
Drug: Binimetinib 15 MG — Binimetinib 15 mg tablet
Drug: Binimetinib 45 MG — Binimetinib 45 mg tablet

SUMMARY:
The current commercially available MEKTOVI® (binimetinib) 15 mg tablets are provided as immediate release film-coated tablets for oral administration. For the treatment of adult patients with unresectable or metastatic melanoma with BRAF V600 mutation, the recommended dosing regimen is 45 mg twice daily (bis in die, BID). No food effect with the commercial formulation of 15 mg was demonstrated. In order to reduce the patient's burden, a new strength tablet containing 45 mg of binimetinib as active ingredient is being developed. As a result, the number of tablets to be taken by the patients will be reduced from 6 tablets (6 x 15 mg) to 2 tablets (2 x 45 mg) per day. The evaluation of the bioequivalence between one 45 mg tablet and three 15 mg tablets is therefore required.

DETAILED DESCRIPTION:
The reference (R) formulation is the currently commercially available tablet containing 15 mg of binimetinib as active substance, administered as three tablets for a total of 45 mg binimetinib. The Test (T) formulation is the tablet containing 45 mg of binimetinib as active substance in one tablet. Participants will be randomized to one of 2 treatment sequences (RT or TR) containing 2 treatment periods, with at least a 7-day washout between each dose.

The study will consist of a screening period between 21 and 2 days before the first study treatment administration on Period (P) 1 Day (D) 1, 2 treatment periods of 5 days each, and a washout of at least 7 days between P1D1 and P2D1.

Study treatments are given by the oral route in fasted condition. The end-of-study (EOS) visit will be performed 30 (± 3) days after the last study treatment administration or discontinuation.

ELIGIBILITY:
Inclusion criteria:

All the following inclusion criteria had to be met for a participant to be eligible to be included in this study:

1. Provide a signed and dated ICF.
2. Healthy participant. Note: defined as an absence of clinically significant abnormalities and any active medical conditions, as identified by a detailed medical history, complete physical examination, vital signs, clinical laboratory tests, cardiac and ophthalmologic evaluation as assessed by the Investigator.
3. Male and female between ≥ 18 and ≤ 65 years of age (at the day of signature of consent).
4. Female participants had to be postmenopausal or sterilized. Note: due to preclinical data of teratogenicity and lack of data on human pregnancies with binimetinib, women of childbearing potential were excluded from this study.

   Women were considered postmenopausal and not of childbearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/mL and estradiol < 20 pg/mL (except if treated with hormone replacement therapy [HRT]) or had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior to dosing. In case of doubt on the menopausal status, the participant was not included. In the case of oophorectomy alone, the reproductive status of the woman was to be confirmed by a follow-up hormone level assessment to consider her of non-childbearing potential.
5. Men with a female partner of childbearing potential were required to use an effective method of birth control or practice abstinence for the entire study duration and for up to 30 days following the last dose of the study treatment.

   Note: the following birth control was recommended: condom for the male participant and an intrauterine device with spermicide or oral or implanted hormonal contraception for the female partner.
6. Body mass index (BMI) of ≥ 18.5 to < 30 kg/m2 with body weight ≥ 50 kg and < 100 kg.
7. Vital signs within the following ranges or if out of normal ranges, considered as not clinically significant by the Investigator except for high diastolic blood pressure (BP): (After at least 5 minutes rest in the supine position)

   1. Supine systolic BP ≥ 90 mmHg and ≤ 140 mmHg
   2. Supine diastolic BP ≥ 50 mmHg and ≤ 90 mmHg
   3. Supine pulse rate (PR) ≥ 45 to ≤ 100 beats per minute (bpm)
   4. Body temperature between ≥ 35.0°C and ≤ 37.5°C
   5. Orthostatic hypotension had to be ruled out based on the following criteria after standing for 5 minutes:

   i. More than a 20 mmHg decrease in systolic BP or 10 mmHg decrease in diastolic BP ii. Clinical signs/symptoms of postural hypotension (dizziness, syncope, etc.), regardless of vital signs.
8. Participants had to have safety laboratory values within the normal ranges or if out of normal ranges considered as not clinically significant by the Investigator except for the following parameters:

   1. Total bilirubin ≤ upper limit of normal (ULN).
   2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyltransferase (GGT) ≤ ULN and alkaline phosphatase (ALP) ≤ 1.1 X ULN.
   3. Serum creatinine within normal range, except on P1D-1 and P2D-1 (≤ 1.1 X ULN).
   4. Serum amylase and lipase ≤ ULN.
   5. Fasting glucose, coagulation panel (prothrombin ratio) within normal range and activated partial thromboplastin time (aPTT) ≤ 1.1 X ULN.

   NB: It was to be noted that for the parameters acceptable at ≤ 1.1 X ULN, if more than one parameter exceeded ULN, the participant was excluded.
9. Able to communicate well with the Investigator and comply with the requirements of the study.
10. Participants had to be willing to comply with dietary and fluid restrictions (from D-7 to 72 hours after the last study treatment administration, see Section 9.4.7.3).
11. Willing to remain in the clinical research unit as required by the protocol.
12. Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.

Exclusion criteria:

Participants meeting any of the following criteria were not eligible to be included in this study:

1. Concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with protocol.
2. Pregnant or currently breastfeeding women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
3. A past medical history of clinically significant ECG abnormalities or a family history (grandparents, parents, and siblings) of prolonged QT interval syndrome.
4. Impaired cardiovascular function.

   Note: including any one of the following:
   1. Left ventricular ejection fraction (LVEF) < 50% or below the institutional lower limit of the normal range (whichever was higher) as determined by standard cardiac echocardiography
   2. Inability to determine the QT interval on ECG
   3. Complete left bundle branch block
   4. Use of a ventricular-paced pacemaker
   5. Congenital long QT syndrome
   6. History of or presence of clinically significant ventricular or atrial tachyarrhythmia
   7. Clinically significant resting bradycardia (< 40 bpm)
   8. History of clinically documented myocardial infarction
   9. History of angina pectoris
   10. History of known structural abnormalities (i.e., cardiomyopathy)
   11. Other clinically significant cardiovascular disease (e.g., congestive heart failure, atherosclerosis, labile hypertension, or uncontrolled hypertension)
   12. Abnormal ECG defined as:

   i. PR interval > 220 msec, QRS complex > 110 msec, QT interval corrected using Fridericia's method (QTcF) > 450 msec (male) and > 470 msec (female) ii. Any ST/T wave abnormalities iii. Any atrial or ventricular arrhythmias, which were of clinical significance and could have had an impact on the safety of the participant or the study as determined by the Investigator iv. Any cardiac conduction abnormalities
5. History of fainting spells or orthostatic hypotension episodes
6. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which might jeopardize the participant in case of participation in the study

   Note: The Investigator was to be guided by evidence of any of the following:
   1. History of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding
   2. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, cholecystectomy or bowel resection
   3. History of, or clinical evidence of, pancreatic injury or pancreatitis
   4. Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests such as ALT, AST, GGT, ALP, or serum bilirubin
   5. Malabsorption syndrome
   6. History of impaired renal function or elevated creatinine values indicating impaired renal function
   7. Evidence of urinary tract obstruction or difficulty in voiding at screening
7. History of autonomic dysfunction or Gilbert syndrome
8. History of immunocompromised status, including a positive human immunodeficiency virus (HIV) infection (enzyme-linked immunosorbent assay and western blot) test result
9. A positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or positive COVID-19 test result or other clinically relevant viral infections
10. Significant illness within the 2 weeks prior to dosing
11. History of clinically significant drug allergy
12. History of atopic allergy (asthma, urticaria, and eczematous dermatitis)
13. Use of any prescription drugs or over-the-counter (OTC) medications (except acetaminophen, i.e., paracetamol) and vitamins, supplements, and herbal remedies within 2 weeks prior to dosing
14. Participants taking acetaminophen (i.e., paracetamol) on a daily basis for more than 2 consecutive days within 1 week prior to dosing was not to be enrolled
15. History or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or ophthalmopathy as assessed by ophthalmologic examination at baseline that would be considered a risk factor for CSR/RVO [e.g., optic disc cupping, visual field defects, intraocular pressure (IOP) > 21 mmHg]
16. Subfoveal choroidal thickness outside of 40μm - 475μm range
17. Neuromuscular disorders that were associated with elevated creatine kinase (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
18. Underwent major surgery ≤ 3 weeks prior to starting study treatment or who had not recovered from side effects of such a procedure
19. Known history or ongoing alcohol abuse within 4 weeks prior to dosing of study treatment Note: alcohol consumption was prohibited 1 week prior to dosing
20. Known regular use of recreational drugs within 4 weeks prior to dosing of study treatment Note: evidence of alcohol abuse/drug use (criterion No. 19 and including this criterion No. 20) as indicated by the laboratory tests conducted during screening or baseline evaluations
21. Smoker or use of tobacco products or products containing nicotine in the 4 weeks prior to first dosing of study treatment Note: smokers were defined as any participant who reported the use of a product containing nicotine during the preceding 30 days or had a positive urine cotinine test > 200 ng/mL
22. Medical, psychiatric, cognitive, or other conditions that could have compromised the participant's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
23. Malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma of the skin (adequate wound healing was required prior to study entry)
    2. Primary malignancy which had been completely resected and was in complete remission for ≥ 5 years
24. History of retinal degenerative disease
25. Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation, or within seven half-lives of the investigational agent taken (whichever was longer) Note: participants who had taken part in a clinical investigation receiving any form of binimetinib had to have completed a 3-week washout prior to baseline
26. Donation or loss of 400 mL or more of blood within 4 weeks prior to dosing
27. Inability to swallow
28. Any vaccination within 4 weeks prior to dosing
29. Participant was under any administrative or legal supervision During the time window authorized for the screening visit (i.e., between 21 and 2 days before admission to the first treatment period), the Investigator could order a re-test of any parameter evaluated during the initial screening visit if he/she needed to evaluate the evolution of said parameter(s) or to confirm the value observed Rechecking of any parameter was to be limited to one time except when the measurement had not been obtained in accurate conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Klein, MD, Principal Investigator — Biotrial
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: No
Pierre Fabre will provide access to individual de-identified data and related study documents [e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)] upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.

RESULTS

PARTICIPANT FLOW:
Groups:
- Binimetinib 45 mg Then Binimetinib 15 mg: Participants first received a single dose of 1 tablet of Binimetinib 45 mg orally in fasted conditions in the morning on day 1 of a five-day period. After a washout period of 7 days, they then received a single dose of 3 tablets of Binimetinib 15 mg orally in fasted conditions in the morning on day 1 of a second five-day period.
Period: Treatment Period 1 (5 Days)
Arm/Group | Binimetinib 15 mg Then Binimetinib 45 mg | Binimetinib 45 mg Then Binimetinib 15 mg
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Binimetinib 15 mg Then Binimetinib 45 mg | Binimetinib 45 mg Then Binimetinib 15 mg
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0
Period: Treatment Period 2 (5 Days)
Arm/Group | Binimetinib 15 mg Then Binimetinib 45 mg | Binimetinib 45 mg Then Binimetinib 15 mg
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Binimetinib 15 mg Then Binimetinib 45 mg | Binimetinib 45 mg Then Binimetinib 15 mg | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (14.05) | 43.9 (13.35) | 42.3 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 19 | 18 | 37
Alcohol history [Count of Participants; unit: Participants]
  Never | 9 | 1 | 10
  Current | 10 | 17 | 27
Smoking history [Count of Participants; unit: Participants]
  Never | 11 | 12 | 23
  Former | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time of Administration to Last Observed Plasma Concentration (AUClast) for Binimetinib
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUClast is defined as area under the concentration from zero to the last quantifiable plasma concentration.
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: The analysis population was the pharmacokinetic set that consisted of 36 healthy participants who had taken one dose of study treatment in the two periods. One participant of the 37 randomised participants was excluded from the pharmacokinetic set due to treatment discontinuation before the second treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Reference Formulation: Binimetinib 3x15 mg
- Test Formulation: Binimetinib 1x45 mg
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h*ng/mL | 1786 (23.22) | 1723 (24.13)
Statistical Analysis 1: Comparison: Reference Formulation vs Test Formulation; Test type: Other; LS-Mean Ratio, Percent = 96.43, 90% CI 2-sided [92.57 to 100.46]

2. Primary Outcome: AUC From Time of Administration to Infinity (AUCinf) for Binimetinib
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUCinf is defined as Area under the plasma concentration-time curve from time of administration to infinity
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h*ng/mL | 1834 (23.09) | 1784 (23.85)
Statistical Analysis 1: Comparison: Reference Formulation vs Test Formulation; Test type: Other; Geometric Mean Ratio = 97.19, 90% CI 2-sided [93.47 to 101.06]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Binimetinib
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Cmax,norm is defined as Cmax divided by dose (mg) per kg body weight.
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
ng/mL | 388.0 (46.3) | 362.2 (41.1)
Statistical Analysis 1: Comparison: Reference Formulation vs Test Formulation; Test type: Other; Geometric Mean Ratio = 94.02, 90% CI 2-sided [87.25 to 101.33]

4. Secondary Outcome: Time to Reach Cmax (Tmax) for Binimetinib
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h | 1.0000 [0.500 to 3.000] | 0.7500 [0.500 to 2.000]

5. Secondary Outcome: Terminal Half-life (t1/2) for Binimetinib
Description: The apparent terminal elimination half-life (t½) is defined as the time necessary for the concentration of a drug to decrease by one-half in the terminal phase
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h | 13.002 (26.194) | 13.901 (24.696)

6. Secondary Outcome: First Order Terminal Elimination Rate Constant (λz) of Binimetinib
Description: The first Order Terminal Elimination Rate Constant (λz) of Binimetinib corresponds to the rate at which a drug is removed from the human system
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
/h | 0.05331 (26.19381) | 0.04986 (24.69575)

7. Secondary Outcome: Residual Area (AUC_%Extrap_obs) for Binimetinib
Description: The residual area under the curve is expressed as a percentage of the total AUC extrapolated from tz to ∞, based on the area under the concentration-time curve.
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of the total AUC
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
% of the total AUC | 2.2836 (53.7862) | 2.8499 (64.4826)

8. Secondary Outcome: Mean Residence Time (MRT) for Binimetinib
Description: Mean residence time (MRT) is defined as the average time for binimetinib to reside in the body
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h | 11.67 (22.66) | 12.588 (27.196)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time of Administration to Last Observed Plasma Concentration (AUClast) for AR00426032
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUClast is defined as area under the concentration from zero to the last quantifiable plasma concentration of AR00426032, a metabolite of binimetinib
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h*ng/mL | 223.9 (29.4) | 213.5 (32.0)

10. Secondary Outcome: AUC From Time of Administration to Infinity (AUCinf) for AR00426032
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUCinf is defined as Area under the plasma concentration-time curve from time of administration to infinity of AR00426032, a metabolite of binimetinib
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 16 | 18
h*ng/mL | 296.8 (18.7) | 287.5 (23.3)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for AR00426032
Description: Cmax is referred as the maximum observed concentration of AR00426032 in blood plasma determined by bioanalysis
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
ng/mL | 41.62 (41.19) | 37.88 (44.25)

12. Secondary Outcome: Time to Reach Cmax (Tmax) for AR00426032
Description: The timepoint at which the maximum concentration of AR00426032 is determined by bioanalysis in the blood plasma
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 36
h | 1.1250 [0.750 to 5.000] | 1.000 [0.750 to 3.000]

13. Secondary Outcome: Terminal Half-life (t1/2) for AR00426032
Description: as for outcome 5
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 16 | 18
h | 13.924 (24.955) | 13.843 (19.281)

14. Secondary Outcome: First Order Terminal Elimination Rate Constant (λz) of AR00426032
Description: The first Order Terminal Elimination Rate Constant (λz) of AR00426032 corresponds to the rate at which a drug is removed from the human system
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 16 | 18
/h | 0.04978 (24.95496) | 0.05007 (19.28093)

15. Secondary Outcome: Mean Residence Time (MRT) for AR00426032
Description: Mean residence time (MRT) is defined as the average time for AR00426032 to reside in the body
Time Frame: Pre-dose = 0h and at 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 16 | 18
h | 14.900 (23.150) | 14.952 (22.934)

16. Secondary Outcome: Clinically Significant Changes From Baseline of Blood Hematology Parameters
Description: Clinically significant shift from baseline in blood hematology parameters (Erythrocytes (red blood cells, RBC), hematocrit, hemoglobin, platelets; leukocyte count with differential: basophils, eosinophils, lymphocytes, monocytes, neutrophils/absolute neutrophil count; RBC indices: mean corpuscular hemoglobin, mean corpuscular volume, reticulocytes/erythrocytes.)
Time Frame: Blood samples for hematology parameters were taken at screening, on Day -1 of each period, at H24 and H48 post-dose of each period, and at end of study (EOS)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

17. Secondary Outcome: Clinically Significant Changes From Baseline of Clinical Chemistry Parameters
Description: Clinically significant shift from baseline in clinical chemistry parameters (alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), bilirubin, gamma glutamyl transferase (GGT), indirect bilirubin, creatinine, urea, bicarbonate, calcium, chloride, magnesium, potassium, sodium, glucose, cholesterol, urate, albumin, creatine kinase (CK), lactate dehydrogenase, protein, amylase, and lipase)
Time Frame: Blood samples for clinical chemistry parameters were taken at screening, on Day -1 of each period, at H24 and H48 post-dose of each period, and at EOS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

18. Secondary Outcome: Clinically Significant Changes From Baseline of Coagulation Parameters
Description: Clinically significant shifts from baseline in coagulation parameters (activated partial thromboplastin time and prothrombin time)
Time Frame: Blood samples for coagulation parameters were taken at screening, on Day -1 of each period, at H24 and H48 post-dose of each period, and at EOS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

19. Secondary Outcome: Clinically Significant Changes From Baseline of Urinalysis Parameters
Description: Clinically significant changes from baseline in the quantitative assessment of pH, bilirubin, erythrocytes, glucose, ketones, leukocyte esterase, nitrite, protein, and urobilinogen
Time Frame: Urinalysis samples were taken at screening, on Day -1 of each period, at H24 and H48 post-dose of each period, and at EOS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

20. Secondary Outcome: Clinically Significant Abnormalities Values of Vital Sign Parameters
Description: Number of participants with at least one clinically significant vital signs abnormality. The following clinical signs were measured: supine and standing systolic and diastolic blood pressure (mmHg), pulse rate (beats/min) body temperature (°C), body weight, and BMI
Time Frame: Vital signs were measured at screening, on Day -1 of each period, at Day 1 pre-dose, H24 and H72 post-dose of each period, and at EOS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

21. Secondary Outcome: Clinically Significant Orthostatic Hypotension
Description: The number and percentage of participants with at least one orthostatic hypotension defined as standing systolic blood pressure (SBP) - supine SBP ≤ -20 mmHg or standing diastolic blood pressure (DBP) - supine DBP ≤ -10 mmHg considered clinically significant.
Time Frame: as for outcome 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 1

22. Secondary Outcome: Clinically Significant Abnormalities Values in 12-lead Electrocardiograms (ECG)
Description: Number of participant with at least one clinically significant electrocardiogram abnormality. The following standard 12-lead ECG parameters were recorded: heart rate (beats/min), PR interval (msec), QRS duration (msec), QRS axis (deg), QT interval (msec) and Fridericia QTc interval (msec)
Time Frame: ECG abnormalities were recorded in triplicate at screening, on Day -1 of each period, at Day 1 pre-dose and H24 post-dose of each period, and at EOS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

23. Secondary Outcome: Clinically Significant Physical Examination Abnormalities
Description: Number of participants with at least one clinically significant physical examination abnormality. A complete physical examination, including at minima assessments of the cardiovascular, dermatological, ear/nose/throat, eyes, gastrointestinal, general health/overall appearance, head, lymph, musculoskeletal, neck, neurological, and respiratory systems was performed
Time Frame: A complete physical examination was performed at screening, on Day -1 of each period, at H24 post-dose of each period, and at EOS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

24. Secondary Outcome: Abnormal Changes From Baseline in Visual Examinations
Description: Visual assessment was performed at screening, on Day -1 of each period, at H24 and H72 post-dose of each period, and at EOS
Time Frame: A visual examination was performed at Screening at at EOS.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 0 | 0

25. Secondary Outcome: Abnormal Changes From Baseline in Ophthalmologic Examinations
Description: Abnormal changes from baseline in ophthalmologic examinations including best corrected visual acuity for distance testing, optical coherence tomography and/or fluorescein angiography, slit lamp examination, IOP and dilated fundoscopy with attention to retinal abnormalities
Time Frame: An opthalmologic examination was performed at Screening at at EOS.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Formulation | Test Formulation
Number analyzed (Participants) | 36 | 37
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time of consent until the end of the follow-up period (up to 30 days after Treatment period 2) and over a total period of 47 days.
Description: AEs were summarized by worst grade according to the NCI-CTCAE V5.0 per participant.
  The analysis population was the safety set that consisted of the healthy participants who had taken one dose of study treatment in the two periods. One participant of the 37 randomised participants discontinued treatment before the second treatment period and therefore did not receive the reference formulation binimetinib 15 mg.
Arm/Group | Reference Formulation | Test Formulation
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 5/36 | 4/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Formulation (N=36) | Test Formulation (N=37)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT05810740/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT05810740/SAP_001.pdf